CLINICAL TRIAL: NCT00379418
Title: Anti Ischemic Effects of Abciximab in Angioplasty and Stenting Patients (AIR)
Brief Title: Anti Ischemic Effects of Abciximab in Angioplasty and Stenting Patients
Acronym: AIR
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kreton Mavromatis, MD, FACC, Assistant Professor, Emory University
Other Study IDs: IRB00021864
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Abciximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Abciximab
  Other Names: Reopro

SUMMARY:
AIR STUDY

TITLE: Anti-Ischemic effects of Abciximab(Reopro)

PATIENT POPULATION: Patients undergoing PCI(an interventional procedure placing a small stent/metallic tube to keep a narrowed artery in your heart open) and either on a stable statin dose or not on a statin. Statin= cholesterol lowering drug(ie, lipitor, zocor).

INTERVENTION: Heparin vs. heparin + abciximab during PCI

PURPOSE: Measure the effects of abciximab on special healing blood stem cells (EPC's-Endothelial Progenitor Cells), on inflammation, on oxidative stress and on microvascular blood flow.

PATIENT ASSESSMENT:

1. 50ccs blood draw on day 1(from sheath), day 2 ,day 7 and day 28.
2. Measurement of blood flow in selected suitable patients
3. 10 minute questionnaire before discharge and on visit on day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Have either:

   * clinical history of anginal symptoms or positive stress test or
   * in stent restenosis
2. Have an angiographic >70% coronary artery stenosis that will be treated with coronary angioplasty or stenting procedure
3. For at least four weeks prior to the procedure have been on, no Hmgcoa- reductase inhibitor or a stable statin dose
4. negative pregnancy test
5. are able to give informed consent

Exclusion Criteria:

1. Coronary intervention within four weeks prior to enrollment.
2. Treatment with abciximab antagonist within four weeks.
3. treatment with thrombolytic therapy within 48 hours
4. MI within 2 months.
5. recent infections
6. general anesthesia within 3 months.
7. renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease undergoing left heart catheterization
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2003-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, M.D., Principal Investigator — EUH
Locations (2):
- United States (2):
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia